CLINICAL TRIAL: NCT05310656
Title: The Effect of Mindfulness Based Empowerment Program on Self-Compassion, Self-Esteem and Ways of Coping With Stress of Women Experienced Violence: A Randomized-Controlled Study
Brief Title: Evaluation of the Impact of the Empowerment Program on Sheltered Battered Women
Acronym: Violence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Elif Güzide Emirza (Other)
Collaborators: Gazi University (Other)
Responsible Party: Sponsor-Investigator, Elif Güzide Emirza, Research Assistant, Gazi University
Organization: Gazi University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: EGUAY
Record Dates: First submitted 2022-03-04; First posted 2022-04-05 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Battered Women; Violence, Domestic; Mindfulness
Keywords: women; violence; mindfulness; empowerment programme; self-compassion

STUDY DESIGN:
Intervention Model Description: The universe of the research will be the women who have been subjected to violence staying in women's shelters in a province in Turkey. Women who volunteer to participate in the study will be included in the study. As a result of the power analysis using the G*Power 3.1 program; With 95% power, 5% margin of error and d=0.84 effect size, a total of at least 42 samples was found to be sufficient (n₁=21; n₂=21). However, considering that losses may also occur, it was planned to work with a total of 60 women, 30 of whom were interventions and 30 were controls. Women who meet the inclusion criteria will be randomly assigned to the intervention and control groups, and at the same time, stratified block randomization will be performed (n₁= 30; n₂=30). The number of people in the group was determined as 10 for reasons such as keeping individuals active, increasing interactive working time, and providing more sharing opportunities.
Masking Description: Due to the nature of the research, it is not possible to blind the researcher and the participant because the researcher applied the mindfulness-based empowerment program, took part in the data collection and analysis phase, and the women in the intervention group were aware of the practice.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindfulness-based empowerment programme (Experimental)
  Interventions: Behavioral: Mindfulness Based Empowerment Programme

INTERVENTIONS:
Behavioral: Mindfulness Based Empowerment Programme — Mindfulness Based Strengthening Program consists of 8 sessions, once a week. Each session has specific goals and objectives, and each session also has a separate theme along with its subject. The subject of the program sessions is as follows: 1st session; Getting to know, explaining the operation plan of the program, defining violence against women and its causes, 2nd session; Emotions and Perceptions, session 3; Being in the Body and Developing Self-Esteem; Session 4, Stress and Meeting Stress with Conscious Awareness; Session 5, The Case of Violence and the Meanings We Ascribe; Session 6, Aware Communication and Conflict Resolution; Session 7, Self-Care and Self-Compassion; Session 8 is Ending the Empowerment Program, Farewell, and a New Beginning. Each session is planned to last an average of 90-120 minutes. Mindfulness teachings and practices will be applied in the content of the program.

SUMMARY:
This study aims to increase the level of self-compassion, improve their self-esteem and cope with stress so that women who are exposed to violence can fight violence more effectively, protect their physical and mental health, find the strength they need to direct their lives, and do all these through self-awareness, compassion and kindness. It is aimed to gain coping skills. For this purpose, a mindfulness-based strengthening program will be implemented.

DETAILED DESCRIPTION:
When the statistics on violence against women in the world are analyzed, it is seen that 16-25% of women are physically abused by their husbands, boyfriends or fiancees, and one out of every five women is exposed to this type of violence in their own home. It has been concluded that the approaches applied in intervention studies for women exposed to violence affect women's mental health positively, increase their self-esteem, improve their coping, problem-solving and decision-making skills, reduce their anger and stress levels, and increase their self-efficacy. In addition, it has been determined that mindfulness-based interventions applied to women who have been subjected to violence strengthen awareness and self-compassion, improve sense of belonging, compassion and problem-solving skills, reduce self-blame, depression, anxiety and suicidal thoughts, increase psychological well-being, and reduce PTSD symptoms. With the continuation of exposure to violence, women are insufficient to change their feelings and lives in a positive way, they are affected by the negative and judgmental attitudes of their environment, they struggle with all the negative effects of violence throughout their lives, they experience physical and mental disorders due to violence, and therefore they resort to harmful coping methods. In this sense, the aim of the study is to determine the effect of mindfulness-based empowerment program on self-compassion, self-esteem and ways of coping with stress in women exposed to violence.

The hypotheses of this study:

In the mindfulness-based empowerment program applied to women who have been subjected to violence, H0-1: There is no difference between the intervention group and the control group in terms of self-compassion.

H0-2: There is no difference between the intervention group and the control group in terms of self-esteem.

H0-3: There is no difference between the intervention group and the control group in terms of coping styles with stress.

ELIGIBILITY:
Inclusion Criteria:

* Women who have been exposed to at least one of the types of violence,
* Women who can read, write and understand Turkish will be included in the study.

Exclusion Criteria:

* Women with severe mental retardation,
* Women with psychotic symptoms and impaired ability to assess reality,
* Women who do not have insight due to psychiatric disorder,
* Women whose cognitive functionality is impaired,
* Women with any physical limitations will not be included in the study.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — The program to be implemented for women who have been subjected to violence aims to strengthen the individual and social empowerment of women who are isolated due to the violence and oppression they are exposed to. Due to violence against women in society, many women have been oppressed and their empowerment has been hindered. For this reason, women who have been traumatized, excluded and subjected to violence are included in the study.
Enrollment: 60 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2022-07-18 (Estimated); Study Completion 2022-08-18 (Estimated)

PRIMARY OUTCOMES:
Self-Esteem | 8 weeks after enrollment
  Coopersmith Self-Esteem Scale: Coopersmith (1967) found the reliability coefficient of the scale to be 0.91 for women and 0.80 for men. In addition, the Cronbach's alpha coefficient of the scale was determined as 0.86. Each item of the scale, which consists of 25 items, is determined according to two options as "suitable for me" and "not suitable for me". Scoring of the scale is made as "4" for each correct statement, "0" for each incorrect statement, the highest score that can be obtained from the scale is 100, and the lowest score is 0. As the score obtained from the scale increases, the self-esteem of individuals also increases. In the scale, a self-esteem level below 50 points is considered low, and a self-esteem level above 50 points is considered high. There is no reverse coded item in the scale.

SECONDARY OUTCOMES:
Ways of Coping with Stress | 8 weeks after enrollment
  Styles of Coping with Stress Scale: The scale consists of 30 items in total. The scale is a 4-point Likert type measurement tool. Options are rated as "Not at all suitable", "Not very suitable", "Appropriate" and "Totally appropriate". In the evaluation of the scale, the total score cannot be obtained, and the scores are calculated separately for each subscale. The answers given to each item are scored as 0,1,2,3, and the scores of each individual in each subgroup are summed up one by one and divided by the number of items in that group. Thus, the average score of each subgroup is obtained. However, items 1 and 9 in the Seeking Social Support group are reverse scored. The increase in the scores obtained from each subscale indicates that the approach of that scale is used more strongly.

OTHER OUTCOMES:
Self-Compassion | 8 weeks after enrollment
  Self-Compassion Scale: The scale is a measurement tool that evaluates the characteristics associated with the sub-dimensions of self-compassion and is based on the individual giving information about himself (self-report). The Self-Compassion Scale has a 5-point Likert-type rating: (1) never (2) rarely (3) often (4) often and (5) always. The scale consists of 26 items. In the confirmatory factor analysis, the existence of 6 sub-dimensions constituting the self-compassion structure was confirmed.

CONTACTS AND LOCATIONS:
Overall Officials: Elif Güzide Emirza, Res. Asist., Principal Investigator — Gazi University

IPD SHARING:
Plan to Share IPD: Yes
It is planned to share the study protocol, data analysis, informed consent form and clinical study report of the study.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: March 2022-December 2022

REFERENCES:
- [Derived] Emirza EG, Bilgili N. The Effect of Mindfulness-Based Empowerment Program on Self-Compassion, Self-Esteem and Ways of Coping With Stress of Women Experienced Violence: A Randomised Controlled Study. Int J Ment Health Nurs. 2024 Dec;33(6):2314-2325. doi: 10.1111/inm.13401. Epub 2024 Aug 12. PMID 39135298